CLINICAL TRIAL: NCT03205215
Title: Hyperbaric Oxygen for Post Concussive Syndrome
Acronym: HBOT for PCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Harrison, Medical Manager and Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H18-01291
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Post-Concussion Syndrome
Keywords: Hyperbaric oxygen; Pressurized oxygen; Concussion; Post concussive syndrome; Oxygen therapy
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): This arm will receive hyperbaric oxygen therapy once consented.
  Interventions: Other: Hyperbaric Oxygen Therapy
- Waitlist - to be treated (Experimental): This arm will receive a hyperbaric oxygen therapy after waiting two months.
  Interventions: Other: Waitlist Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — 100% oxygen delivered by hood at 2 ATA for 90 minutes with 5 minute air breaks
  Arms: Immediate Treatment
Other: Waitlist Hyperbaric Oxygen Therapy — 100% oxygen delivered by hood at 2 ATA for 90 minutes with 5 minute air breaks
  Arms: Waitlist - to be treated

SUMMARY:
We would like to see if Hyperbaric Oxygen can help improve the symptoms that result from Post Concussive Syndrome.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to examine the role of Hyperbaric Oxygen Therapy (HBOT) in decreasing symptoms in patients with a diagnosis of chronic post concussive syndrome (PCS).

Hypothesis:

The study hypothesis is that HBOT will decrease symptoms measured by standard measurement tools when provided to patients who have a diagnosis of PCS and are 6 months to 36 months post injury.

Study Overview:

Hyperbaric oxygen therapy (HBOT) involves the administration of inhaled 100% oxygen at increased ambient pressure inside a closed vessel. HBOT produces greatly elevated arterial and tissue oxygen tensions, producing a wide variety of physiological effects at the cellular and sub cellular level.

Participants will be selected from the post-concussive syndrome population based on an expectation that they would experience a clinically significant improvement. Eligible subjects will be experiencing post concussive symptoms related to an injury within the last 6 to 36 months. The study will be enrolling 150 participants and will be randomized to two different treatment arms: experimental group and a waitlist group.

Each participant will receive a series of forty 2 hour treatments, delivered once a day, 5 days a week, within the hyperbaric oxygen chamber.There will be assessments completed before treatment series begins, at the end of treatment, 8 months and 14 months after treatment begins. The primary outcome will be administered at these times as well as every two weeks once treatment begins until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak English and give informed consent.
* A diagnosis of chronic PCS made by a referring physician
* Time of injury between 6 and 36 months previously
* Able to sit in the chamber for 120 minutes.

Exclusion Criteria:

* Untreated collapsed lung (pneumothorax)
* Have taken the chemotherapy drug Doxorubicin within 72 hours
* Have taken the chemotherapy drug Bleomycin within 4 months
* Bowel obstruction
* Heart pacemaker that has not been certified as safe for exposure to 2.0 ATA
* Pregnancy
* Severe Chronic Obstructive Pulmonary Disease (COPD)
* Participation in other PCS related studies.
* Previous recent HBOT
* Previous recent deep sea diving experience

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Rivermead Post Concussion Syndrome Questionnaire | Baseline, after 10, 20, 30 hyperbaric treatments, 2, 2.5, 3, 3.5, 4,4.5, 5, 5.5 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5 and 14 months post baseline,
  15 questions regarding a participant's Post Concussive symptoms

SECONDARY OUTCOMES:
Change in the NIH Tool Box | Baseline, 2 months post baseline, 8 months post baseline, 14 months post baseline
  Cognitive Assessment Cluster
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 2 months post baseline, 8 months post baseline, 14 months post baseline
  Depression Assessment
Change in the Short Form Health Survey (SF-36) | Baseline, 2 months post baseline, 8 months post baseline, 14 months post baseline
  Quality of Life Assessment
Change in the Quality of Life After Brain Injury (QOLIBRI) | Baseline, 2 months post baseline, 8 months post baseline, 14 months post baseline
  Quality of Life Assessment
Change in the WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline, 2 months post baseline, 8 months post baseline, 14 months post baseline
  Daily Functioning Assessment

CONTACTS AND LOCATIONS:
Overall Officials: David W Harrison, MD,CCFP(EM),FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital - Hyperbaric Unit, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No